CLINICAL TRIAL: NCT05040906
Title: A Phase 3, Randomized, Double-blind Study of H02 Plus CHOP Versus R-CHOP in Patients With Diffuse Large B-cell Lymphoma
Brief Title: A Study Comparing the Efficacy and Safety Between H-CHOP and R-CHOP in Untreated CD20-Positive Diffuse Large B-cell Lymphoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTP-H02-Ⅰ-Ⅲ
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Recruiting
Keywords: DLBCL; CD20; R-CHOP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H02+ Chemotherapy (Experimental): Participants received six cycles of H02(375 mg/m2) combined with six cycles of standard cyclophosphamide,doxorubicin,vincristine,and prednisone/prednisolone(CHOP) chemotherapy(21-day cycles).
  Interventions: Drug: H02+CHOP
- Rituxan+Chemotherapy (Active Comparator): Participants received six cycles of Rituxan combined with six cycles of standard cyclophosphamide,doxorubicin,vincristine,and prednisone(CHOP) chemotherapy(21-day cycles).
  Interventions: Drug: Rituxan +CHOP

INTERVENTIONS:
Drug: H02+CHOP — Drug:H02 375 mg/m2,administered intravenously(IV) on Day1 of each 21-day cycle for 6 cycles.
  Drug : Cyclophosphamide 750 mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug:Doxorubicin 50 mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Vincristine 1.4mg mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Prednisone 100 mg administered orally on Days 2-6 of each 21-day cycle.
  Arms: H02+ Chemotherapy
Drug: Rituxan +CHOP — Drug: Rituxan 375 mg/m2,administered intravenously(IV) on Day1 of each 21-day cycle for 6 cycles.
  Drug : Cyclophosphamide 750 mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Doxorubicin 50 mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug : Vincristine 1.4mg mg/m2,administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Prednisone 100 mg administered orally on Days 2-6 of each 21-day cycle.
  Arms: Rituxan+Chemotherapy

SUMMARY:
This trial is a Multicenter, randomized, double-blind, parallel, controlled, and equivalence phase Ⅲ study.

Primary objective:

The purpose is to compare the objective response rate of H02 (rituximab biosimilar) plus CHOP and rituximab plus CHOP, as first-line treatment of diffuse large B-cell lymphoma.

Secondary objective:

The purpose is to compare the safety of H02 combined with CHOP regimen and rituximab injection (Rituximab®) combined with CHOP regimen in the treatment of newly treated diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated CD20-positive DLBCL confirmed.
2. 18 years to 75 years; Male or female patients.
3. IPI score of 1 to 2 and an ECOG performance status of 0 to 2.
4. More than 6 months life expectancy.
5. At least one measurable lymph node:
6. For intranodal lesions, equal or greater than 1.5 cm in the long axis and equal or greater than 1.0 cm in the short diameter; For extranodal lesions, equal or greater than 1.0 cm in the long axis.
7. Adequate cardiac function (LVEF≥50%).
8. Absolute neutrophil count(ANC) ≥1.5*109/L and platelet count(PLT) ≥75*109/L and hemoglobin ≥75g/L, total bilirubin level ≤1.5×upper limit of normal (ULN), aspartic acid Aminotransferase (AST), alanine aminotransferase (ALT)≤2.5×ULN, creatinine level (Cr)≤1.5×ULN.
9. Signed an informed consent form which was approved by the institutional review board of the respective medical center.

Exclusion Criteria

1. Primary central nervous system(CNS) lymphoma, secondary CNS involvement, primary skin DLBCL (leg type), primary mediastinal (thymic) large B-cell lymphoma, intravascular large B-cell lymphoma, and primary exudation Lymphoma, T-cell/histiocytosis-rich large B-cell lymphoma, ALK-positive large B-cell lymphoma, plasmablastic lymphoma, lymphoma-like granuloma, EBV-positive mucosal skin ulcer, HHV8+DLBCL, NOS, primary testicular lymphomas.
2. High-grade B-cell lymphoma with MYC, BCL2 and/or BCL6 rearrangement diagnosed by fluorescence in situ hybridization (FISH).
3. B-cell lymphoma has characteristics between DLBCL and classic HL, and cannot be divided into types.
4. Transformed lymphoma. those who have transformed from other types of lymphomas, such as follicular lymphoma, marginal zone B-cell lymphoma, and chronic lymphocytic leukemia/small B-cell lymphoma.
5. History of other malignancy, except for skin basal cell carcinoma and cervical carcinoma in situ and has been in remission without treatment for >/= 5 years prior to enrolment.
6. Severe mental illness.
7. Positive for HIV infection.
8. Positive for HCV infection.
9. Patients who have HBV (+) are eligible.
10. History of anti-CD20 monoclonal antibody treatment for other disease (e.g., rheumatoid arthritis).
11. Previous treatment for NHL, including chemotherapy, immunotherapy, radiotherapy, monoclonal antibody therapy or surgical treatment (except lymph node biopsies diagnostic surgery and biopsy).
12. Participation in another clinical trial in the past 3 months.
13. Vaccination with a attenuated live vaccine within 4 weeks.
14. Use of hemopoietic cytokine in the past 2 weeks, e.g. granulocyte colony stimulating factor(G-CSF).
15. Disease or symptom by the investigator's discretion(interstitial pneumonia, Uncontrollable systemic infections,severe cardiovascular disease (New York Heart Association functional class III or IV, myocardial infarction or unstable arrhythmia or unstable angina in the last 6 months, severe cardiac insufficiency, rogressive multifocal leukoencephalopathy), uncontrolled hypertension (SBP≥180mmHg and/or DBP≥100mmHg), active autoimmune diseases)
16. Known hypersensitivity to any of the study drugs or its ingredients.
17. Prior treatment with anthracycline.
18. DLBCL invaded by special parts such as testis, breast, ovary, etc.
19. Pregnant or lactating women.
20. The researcher believes that it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(based on the evaluation of the IRC) | 18 weeks
  To evaluate the objective response rate (ORR) in patients with previously untreated Diffuse Large B-cell Lymphoma after six periods of treatment.

SECONDARY OUTCOMES:
ORR(based on the judgment of the investigator) | 18 weeks
Complete response (CR) rate (based on the evaluation of the IRC and investigator) | 18 weeks
  CR was defined as the complete disappearance of all previously detectable disease signs. CR rate was percentage of participants with a CR event.
1-year progression-free survival (PFS) rate | 1 year
  PFS was defined as the time from randomization to first occurrence of disease progression, relapse, or death from any cause. The proportion of subjects without disease progression or death from any cause after randomization for one year.
Duration of remission within 1 year (DOR) | 1 year
  The time from the first assessment of complete response or partial response to the first assessment of PD or death after randomization within 1 year.
1-year overall survival (OS) rate | 1 year
  The proportion of subjects who did not die from any cause after randomization for 1 year.
1-year event-free survival (EFS) rate | 1 year
  OS was defined as the time from randomization to death from any cause. Percentage of subjects without disease progression, death, or any interruption of treatment at 1 year of randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong New Time Pharmaceutical Co., LTD, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided